CLINICAL TRIAL: NCT00198081
Title: A Phase II Trial of Celecoxib in Patients With IPMN
Brief Title: Use of Celecoxib in Patients With Intraductal Papillary Mucinous Neoplasms (IPMNs)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding and personnel to conduct study.
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0305-20
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Pancreas Neoplasms
Keywords: celecoxib for pancreas lesions
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cyclooxygenase 2 Inhibitors; Celecoxib; Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgical Candidate (Experimental): COX-2 Inhibitor 6-8 weeks prior to surgery
  Interventions: Drug: COX-2 Inhibitor 6-8 weeks prior to surgery
- Medical Candidate (Experimental): COX-2 Inhibitor for 6 months prior to follow-up EUS or ERCP
  Interventions: Drug: COX-2 Inhibitor for 6 months prior to follow-up EUS or ERCP

INTERVENTIONS:
Drug: COX-2 Inhibitor 6-8 weeks prior to surgery — 400 mg BID 6-8 weeks prior to surgery
  Other Names: Celecoxib
  Arms: Surgical Candidate
Drug: COX-2 Inhibitor for 6 months prior to follow-up EUS or ERCP — 400 mg BID for 6 months prior to follow-up EUS or ERCP
  Other Names: Celecoxib
  Arms: Medical Candidate

SUMMARY:
The purpose of the study is to find out whether the drug celecoxib has beneficial effects on people with pre-cancerous lesions of the pancreas.

DETAILED DESCRIPTION:
Efforts at finding a successful chemotherapy for pancreatic cancer have been disappointing. Some patients are at increased risk of pancreatic cancer or may have pre-malignant pancreatic lesions which predispose them to later pancreatic cancer development. In these individuals, chemopreventative measures may block future development of pancreatic cancer. Human tissue studies, cell culture and animal models of pancreatic cancer strongly suggests that cyclooxygenase-2 (COX-2) may be a successful target for chemoprevention. COX-2 is overexpressed in human pancreatic cancers. Elevated COX-2 expression correlates with progression of premalignant precursors of pancreatic cancer in development models of hamster pancreatic cancer. Human tissue studies confirm increases in COX-2 expression with progression of premalignant precursors called intraductal papillary mucinous neoplasms (IPMNs) and pancreatic intraepithelial neoplasms (PanINs). Moreover, COX-2 inhibitors appear to have chemopreventative efficacy in the PC-1 homograft model of hamster pancreatic cancer. Demographic studies have suggested COX-2 inhibitors may confer protection from pancreatic cancer. We propose to conduct a pilot/phase II trial to determine the chemopreventative effects of the COX-2 inhibitor celecoxib in patients with premalignant pancreatic lesions.

Patients registered to the study will take celecoxib twice daily for 6-8 weeks prior to surgery (if patient decides to have surgery for his/her condition). If subject is not a surgical candidate or puts off surgical treatment, subject will take celecoxib for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of IPMN
* ECOG Performance status of 0, 1, or 2
* Adequate liver function, bilirubin < 1.5 times ULN, ALT or AST < 2.5 times ULN
* Adequate renal function: creatinine < 1.8
* Must be at least 18

Exclusion Criteria:

* Use of COX-2 selective inhibitors within the last month
* More than occasional use of NSAIDS in last month (occasional use defined as up to twice weekly dosing)
* CA19-9 levels 1.5 times the ULN
* Active pancreatitis
* Taking sulphonylureas, fluconazole or lithium concomitantly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian M. Schmidt, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Surgical Candidate | Medical Candidate
Started | 5 (Eight (8) persons consented to participate but 3 withdrew prior to beginning protocol treatment.) | 0 (No enrollment on this arm.)
Completed | 4 | 0 (No enrollment on this arm.)
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Surgical Candidate | Medical Candidate | Total
Number analyzed (Participants) | 5 | 0 | 5
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 2 |  | 2
  >=65 years | 3 |  | 3
Gender [Number; unit: participants]
  Female | 0 |  | 0
  Male | 5 |  | 5
Ethnicity (NIH/OMB) [Number; unit: participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 5 |  | 5
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 1 |  | 1
  Black or African American | 0 |  | 0
  White | 4 |  | 4
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 |  | 5
IPMN type [Number; unit: participants]
  Adenoma | 1 |  | 1
  Low grade | 1 |  | 1
  Invasive | 1 |  | 1
  Not Otherwise Specified | 1 |  | 1
  Unknown | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Concentration of PGE2 in Urine at Baseline, Surgery, 1 wk, 4wks, and 6 Months
Description: Measured by Elisa at participant level - only participant level data available; not summarized across group
Time Frame: Baseline, surgery, 1 wk, 4 wks, and 6 months
Measure: Number; unit: pg/ml
Groups:
- Surgical Candidate Baseline; Surgery Candidate Surgery; Surgical Candidate One Week; Surgical Candidate 4 Weeks; Surgical Candidate 6 Months: COX-2 Inhibitor 6-8 weeks prior to surgery
  COX-2 Inhibitor 6-8 weeks prior to surgery: 400 mg BID 6-8 weeks prior to surgery
Arm/Group | Surgical Candidate Baseline | Surgery Candidate Surgery | Surgical Candidate One Week | Surgical Candidate 4 Weeks | Surgical Candidate 6 Months
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
pg/ml
  IPMN Adenoma-Part 1 | 11800 | 13300 | 12100 | 19600 | 24000
  IPMN low-Part 2 | 21000 | 13400 | 4700 | 36300 | 16000
  IPMN Invasive-Part 3 | 800 | 30000 | 15400 | 24800 | 3600
  IPMN NOS-Part 4 | 10100 | 8700 | 9500 | 40300 | 7500

2. Secondary Outcome: Number of Participants With Clinical Changes in IPMN Progression.
Description: Examine the short term effect of celecoxib on clinical progression of IPMN in the surgical arm; Examine the long term effect of celecoxib on clinical progression of IPMN in the medical arm.
Time Frame: Baseline, 6 months, 1 year
Population: Data never collected for surgical arm; medical arm of study never initiated.
Arm/Group | Surgical Candidate | Medical Candidate
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Concentration of PGE2 in Serum at Baseline, Surgery, 1 wk, 4wks, and 6 Months
Description: Measured by Elisa at participant level - only participant level data available; not summarized across group
Time Frame: Baseline, surgery, 1 wk, 4 wks, and 6 months
Measure: Number; unit: pg/ml
Arm/Group | Surgical Candidate Baseline | Surgery Candidate Surgery | Surgical Candidate One Week | Surgical Candidate 4 Weeks | Surgical Candidate 6 Months
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
pg/ml
  IPMN Adenoma-Part 1 | 60 | 70 | 70 | 130 | 100
  IPMN low-Part 2 | 170 | 90 | 10 | 40 | 10
  IPMN Invasive-Part 3 | 70 | 30 | 60 | 10 | 70
  IPMN NOS-Part 4 | 100 | 140 | 20 | 80 | 30

4. Primary Outcome: Concentration of PGEM in Urine at Baseline, Surgery, 1 wk, 4wks, and 6 Months
Description: Measured by Elisa at participant level - only participant level data available; not summarized across group
Time Frame: Baseline, surgery, 1 wk, 4 wks, and 6 months
Measure: Number; unit: pg/ml
Arm/Group | Surgical Candidate Baseline | Surgery Candidate Surgery | Surgical Candidate One Week | Surgical Candidate 4 Weeks | Surgical Candidate 6 Months
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
pg/ml
  IPMN Adenoma-Part 1 | 196 | 177 | 354 | 431 | 522
  IPMN low-Part 2 | 257 | 201 | 153 | 594 | 366
  IPMN Invasive-Part 3 | 128 | NA — Above the level of detection | 850 | 453 | 184
  IPMN NOS-Part 4 | 131 | 100 | 184 | 417 | 88

5. Primary Outcome: Concentration of PGEM in Serum at Baseline, Surgery, 1 wk, 4wks, and 6 Months
Description: Measured by Elisa at participant level - only participant level data available; not summarized across group
Time Frame: Baseline, surgery, 1 wk, 4 wks, and 6 months
Measure: Number; unit: pg/ml
Arm/Group | Surgical Candidate Baseline | Surgery Candidate Surgery | Surgical Candidate One Week | Surgical Candidate 4 Weeks | Surgical Candidate 6 Months
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
pg/ml
  IPMN Adenoma-Part 1 | 20 | 4 | 6.4 | 5.4 | 6.7
  IPMN low-Part 2 | 7 | 4.3 | 9.3 | 5.9 | 8.7
  IPMN Invasive-Part 3 | 2 | 3 | 11.8 | 5.1 | 8.3
  IPMN NOS-Part 4 | 9 | 3.4 | 7.2 | 4.3 | 1.8

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Surgical Candidate | Medical Candidate
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/0
Other Adverse Events (participants affected / at risk) | 5/5 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgical Candidate (N=5) | Medical Candidate (N=0)
NERVOUS SYSTEM DISORDERS - OTHER, [NEUROLEPTIC REACTION] (Nervous system disorders) | 1 (1) | 0
CARDIAC DISORDERS - OTHER, [CONGESTIVE HEART FAILURE] (Cardiac disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgical Candidate (N=5) | Medical Candidate (N=0)
EKG CHANGES (Cardiac disorders) | 1 (1) | 0
PALPITATIONS (Cardiac disorders) | 1 (1) | 0
ARRTHYTHMIA (Cardiac disorders) | 1 (1) | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0
DIARRHEA (Gastrointestinal disorders) | 2 (2) | 0
PANCREATIC FISTULA (Gastrointestinal disorders) | 1 (1) | 0
PAIN (Gastrointestinal disorders) | 1 (1) | 0
FATIGUE (General disorders) | 2 (2) | 0
EDEMA: LIMB SWELLING OF THE ARMS AND/OR LEGS (General disorders) | 1 (1) | 0
FLU-TYPE SYMPTOMS (INCLUDING BODY ACHES, FEVER, CHILLS, TIREDNESS,LOSS OF APPETITE, COUGH) (General disorders) | 1 (1) | 0
TOOTH INFECTION (Infections and infestations) | 1 (1) | 0
SEROMA (Injury, poisoning and procedural complications) | 1 (1) | 0
INR INCREASED (Investigations) | 1 (1) | 0
PLATELET COUNT DECREASED (Investigations) | 1 (1) | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, [RUNNY NOSE] (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
HYPOTENSION (Vascular disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes